CLINICAL TRIAL: NCT00309400
Title: The Early History of Universal Screening for Metabolic Disorders
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeffrey P. Brosco, Professor, Clinical Pediatrics, University of Miami
Other Study IDs: 20057601
Record Dates: First submitted 2006-03-30; First posted 2006-03-31 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Phenylketonuria; Galactosemia; Inborn Errors of Metabolism
Keywords: History; Phenylketonuria; Galactosemia; Screening; Treatment
MeSH Terms: conditions — Phenylketonurias; Galactosemias; Metabolism, Inborn Errors

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We are doing this study to learn more about the early history of universal screening for metabolic disorders such as PKU and galactosemia. In particular, we are interested in learning from our past experience to inform our current plans to expand universal newborn screening. Following standard historical research methodology, we will begin with a review of the historical scholarship on PKU and galactosemia, including more general works on mental retardation, genetics, public health screening, and metabolic disorders. We will also obtain scientific publications and archival sources on the early screening and treatment of these disorders. Lastly, we will conduct oral history interviews with key participants in teh early screening and treatment of PKU and galactosemia.

DETAILED DESCRIPTION:
Universal neonatal screening programs for metabolic disorders constitute a triumph of medicine and public policy in the US over the last 50 years. State programs to identify and treat disorders such as and galactosemia have saved thousands of lives and prevented serious morbidity such hypothyroidism, phenylketonuria (PKU), as mental retardation . Advances in science and technology, including the Human Genome Project, offer the opportunity to expand universal newborn screening programs to include many new conditions. Although the benefits of such screening programs appear to outweigh their costs, some critics have pointed to historical examples that should make us wary of expanding universal newborn screening. For example, ethicist Norm Fost has stated that early screening programs falsely identified hundreds of children as having PKU or galactosemia, and that inappropriate treatment of these children led to death or severe neurodevelopmental impairment . As our nation weighs the risks and benefits of expanding newborn screening to a variety of metabolic and genetic conditions, it is critical to revisit the early years of universal screening programs. Did the extension of screening from at-risk populations to all newborns lead to substantial morbidity and mortality? If so, what can we learn from our past experience to inform our current plans to expand universal newborn screening?

We propose to examine the early history of universal screening for PKU and galactosemia in the US. Following standard historical research methodology, we will begin with a review of the historical scholarship on PKU and galactosemia, including more general works on mental retardation, genetics, public health screening, and metabolic disorders. We will also identify and obtain scientific publications and archival sources that document the early screening and treatment of these disorders. Lastly, we will conduct oral history interviews with key participants in the history of early screening and treatment of PKU and galactosemia. Oral history is a critical component of this project, providing information not available in any other format. Through oral history interviews, we hope to identify critical events, key people, and important collateral influencing issues.

The second phase of historical methods requires the scholar to identify key themes based on the historical record, then present preliminary findings to groups of scholars from a variety of disciplines. This academic exchange leads the PI to new resources and to refined key themes. The final phase of historical scholarship is preparation of written conclusions. As a result of this project, a historical article will be written for a peer-reviewed journal accessible to clinicians, researchers, and policy experts who are considering how best to expand universal metabolic screening.

ELIGIBILITY:
Inclusion Criteria:

* participants in the history of early screening and treatment of PKU and galactosemia

Exclusion Criteria:

* those who decline to be interviewed

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physicians and scientists knowledgeable about history of newborn screening
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Historical report of PKU false positive morbidity/morality | After newborn screening began (1960)
  This study involved oral history interviews, so outcomes are qualitative

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey P Brosco, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Mailman Center for Child Development, Miami, Florida, United States